CLINICAL TRIAL: NCT01426776
Title: Effect of Heart Valve Replacement on Cheyne-Stokes Respiration in Patients With Rheumatic Heart Disease
Brief Title: Effect of Heart Valve Replacement on Cheyne-Stokes Respiration
Acronym: CSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhang Xilong, Department of Respirology, The First Affiliated Hospital of Nanjing Medical University, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 30971319; 20092801 (Other: Ethic committee)
Record Dates: First submitted 2011-08-28; First posted 2011-08-31 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Cheyne-Stokes Respiration; Heart Valve Disease; Central Sleep Apnea
Keywords: Cheyne-Stokes respiration; Heart valve disease; Central Sleep Apnea
MeSH Terms: conditions — Cheyne-Stokes Respiration; Heart Valve Diseases; Sleep Apnea, Central | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- heart valve replacement (Other): a normal surgery that rheumatic valvular heart disease patients received.
  Interventions: Procedure: heart valve replacement

INTERVENTIONS:
Procedure: heart valve replacement — The patients with heart valve disease and CSR will be received heart valve replacement
  Other Names: cardiac surgery

SUMMARY:
Sleep disordered breathing, especially central sleep apnea, is common in patients with chronic heart failure. Heart valve replacement could have some effect on central sleep apnea. The aim of the study is to investigate effect of heart valve replacement on Cheyne-Stokes respiration in patients with rheumatic heart disease.

DETAILED DESCRIPTION:
Sleep apnea, especially central sleep apnea, has a high prevalence in patients with chronic heart failure. Although sleep disordered breathing (SDB) have been described in patients with heart disease, the prevalence is not known because: ①There are various forms of SDBs, including obstructive sleep apnea(OSA), central sleep apnea (CSA), and mixed forms of sleep apnea syndromes that have variable prevalence; ②Patients suffering from rheumatic valve disease usually have varying degrees of heart failure, and this variability affects estimates of prevalence; ③There are no international patient registries and SDB is underdiagnosed in many parts of the world.

The previous studies are most focusing on nonvalvular disease. We ①investigate the prevalence and the risk factors of Cheyne-Stokes respiration in patients with heart valve diseases, ②compare the changes of parameters of Cheyne-Stokes Respiration and heart function (like apnea hypopnea index, pulse oxygen saturation, blood pressure, echocardiogram, electrocardiogram, 6-minute walk test) before heart valve replacement and 3, 6, and 12 months after the surgery.

With nocturnal polysomnography (PSG) examination 30 patients typical CSR are going to be screened out from 300 patients with heart valve disease and waiting for cardiac surgery. The Comparison of 30 patients undergoing heart valve replacement will be performed before and 3, 6, and 12 months following heart valve replacement. We shall analyze the changes of CSR before and after valve replacement as well as the correlation among cardiac function and PSG parameters.

ELIGIBILITY:
Inclusion Criteria:

* heart valve disease with any ejection fraction
* clinical diagnosis of Cheyne-Stokes respiration

Exclusion Criteria:

* unstable heart failure
* stroke
* transient ischemic attack in last 6 months
* pacemaker, cardioverter-defibrillator or resynchronization device implanted less than 6 months before study entrance
* severe chronic obstructive pulmonary disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Changes of CSR index before and 3, 6, 12 months following valve replacement. | 1 year after cardiac surgery of each enrolled patient
  The primary goal of this study is to compare the changes of polysomnography(PSG) parameters(index of CSR, apnea hypopnea index, pulse oxygen saturation, etc)before and 3, 6, 12 months following the cardiac valve replacement surgery.

SECONDARY OUTCOMES:
Association of PSG parameters with cardiac function before and 3, 6, 12 months following valve replacement | 1 year after cardiac surgery of each enrolled patient
  The secondary goal of this study is to determine the association of PSG parameters(index of CSR, apnea hypopnea index, pulse oxygen saturation, electrocardiogram, etc)and cardiac function (LVEF, 6-minute walk test, etc) before and 3, 6, 12 months following the cardiac valve replacement surgery. Qualities of life and sleep will also be masured before and 3, 6, 12 months after surgery. (The quality of life is assessed by reference to "The Medical Outcomes Study 36item Short-Form Health Survey"(SF-36) generic questionnaire, and sleep quality is assessed by Pittsburgh Sleep Quality Index(PSQI).)

CONTACTS AND LOCATIONS:
Overall Officials: Shijiang Zhang, MD, Study Director — The First Affiliated Hospital with Nanjing Medical University; Ning Ding, Doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Abe H, Takahashi M, Yaegashi H, Eda S, Kitahara H, Tsunemoto H, Kamikozawa M, Koyama J, Yamazaki K, Ikeda U. Valve repair improves central sleep apnea in heart failure patients with valvular heart diseases. Circ J. 2009 Nov;73(11):2148-53. doi: 10.1253/circj.cj-09-0307. Epub 2009 Aug 28. PMID 19713650
- [Result] Rubin AE, Gottlieb SH, Gold AR, Schwartz AR, Smith PL. Elimination of central sleep apnoea by mitral valvuloplasty: the role of feedback delay in periodic breathing. Thorax. 2004 Feb;59(2):174-6. doi: 10.1136/thorax.2003.007799. PMID 14760162
- Available data/document: published article: PMID: 24938583 — https://pubmed.ncbi.nlm.nih.gov/24938583 — We found central sleep apnea was eliminated after cardiac valve replacement surgery, however, there was no change in obstructive sleep apnea.